CLINICAL TRIAL: NCT06545812
Title: Serum Concentrations of Cytokines and Metallopeptidases During the Conservative and Minimal Invasive Treatment of Pain Caused by Lumbar Disc Herniation
Brief Title: Immune Response During the Conservative and Minimal Invasive Treatment of Pain Caused by Lumbar Disc Herniation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Josip Juraj Strossmayer University of Osijek (Other)
Responsible Party: Principal Investigator, Karla Rožac, researcher in the doctoral study of Molecular Biosciences, Faculty of dental medicine and health Osijek, Josip Juraj Strossmayer University of Osijek
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2158/97-97-10-24-50
Record Dates: First submitted 2024-07-23; First posted 2024-08-09 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Intervertebral Disc Herniation; Back Pain; Analgesic Nephropathy; Inflammatory Response
Keywords: Bulging of intervertebral disc;; Physical therapy;; Epidural steroid injection (ESI);; Pro-inflammatory cytokines;; Anti-inflammatory cytokines;; Metallopeptidases;
MeSH Terms: conditions — Intervertebral Disc Displacement; Back Pain | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical therapy for disc herniation (Active Comparator): Conservative treatment in the form of physical therapy consists of several physical factors, namely laser therapy, ultrasound and transcutaneous electroneurostimulation (TENS). Blood samples for analysis for multicomplex quantitative analysis of anti-inflammatory cytokines (interleukin 1β (IL-1β), interleukin 6 (IL-6), interleukin 8 (IL-8), interferon gamma (INF-γ), tumor necrosis factor alpha or gamma (TNF-α), chemokine ligand 3 (CCL3) and matrix metalloproteinases MMP-3 and MMP-9
  Interventions: Device: Physical therapy for disc herniation
- Epidural steroid injection (ESI) (Active Comparator): Minimally invasive methods such as epidural steroid injection (ESI). Blood samples for analysis for multicomplex quantitative analysis of anti-inflammatory cytokines (interleukin 1β (IL-1β), interleukin 6 (IL-6), interleukin 8 (IL-8), interferon gamma (INF-γ), tumor necrosis factor alpha or gamma (TNF-α), chemokine ligand 3 (CCL3) and matrix metalloproteinases MMP-3 and MMP-9
  Interventions: Drug: Transforaminal epidural steroid injection

INTERVENTIONS:
Drug: Transforaminal epidural steroid injection — Transforaminal epidural steroid injection (ESI TF) with corticosteroids like Methylprednisolone, Levobupivacaine and Lidocaine according to the protocol of the institution. They reduce inflammation by inhibiting pro-inflammatory mediators and causing a reversible local anesthetic effect.
  Other Names: ESI TF
  Arms: Epidural steroid injection (ESI)
Device: Physical therapy for disc herniation — BTL Laser therapy, BTL ultrasound therapy and BTL Transcutaneous electrical nerve stimulation - TENS
  Arms: Physical therapy for disc herniation

SUMMARY:
Bulging of the intervertebral disc in the lumbar part of the spine is one of the most common degenerative changes of the spine in the elderly population, which causes various symptoms such as radicular pain. Possible mechanisms of radicular pain are mechanical compression of the intervertebral disc on the nerve and sterile local inflammation caused by proinflammatory factors. Depending on the degree of diagnosis, if conservative treatment is not successful, then treatment is focused on minimally invasive methods such as epidural steroid injection (ESI). The achieved neural blockade is believed to alter or interrupt nociceptive input, reflex mechanisms induced by afferent fibers, self-sustaining neuronal activity, and central neuronal activity. On the other hand, corticosteroids reduce inflammation by inhibiting pro-inflammatory mediators and causing a reversible local anesthetic effect. The aim of the research is to measure the concentrations of pro-inflammatory and anti-inflammatory cytokines and metallopeptidases in the serum before physical therapy, i.e. ESI, and two weeks and three months after the start of said therapies, then to examine the clinical status, intensity of pain and limitations of movement associated with pain in all three time points in order to determine the treatment outcomes after the mentioned therapies and examine the possible association of cytokine concentrations with the treatment outcomes and, last but not least, to determine the degree of the patient's psychophysical condition and quality of life before the mentioned therapies, two weeks and three months after the start of the therapies in order to examined possible associations with treatment outcomes and changes in cytokine and metallopeptidases concentrations.

DETAILED DESCRIPTION:
The location of the research is the Institute for Pain Management at the Clinic for Anesthesiology, Reanimatology and Intensive Care, Clinical Hospital Center Osijek, then the Translational Medicine Laboratory of the Faculty of Dental Medicine and Health Osijek. The research is designed as a non-randomized controlled experiment, and the duration of the research will depend on the available number of patients who meet the inclusion criteria for the mentioned research, and considering the expected influx of patients, the planned duration is 18 months.

All patients will receive written informed consent and the procedure will be explained orally. After signing the informed consent, the patients will be divided into two groups. One group of patients will undergo epidural administration of steroids and local anesthetic through a transforaminal approach, and the other group of patients will undergo a conservative pain management method. All subjects will be selected at the Institute for Pain Management of KBC Osijek. Below are the criteria for inclusion and exclusion of patients in this study.

By inspecting the medical documentation, all the ethical and moral rights of the respondents will be respected, with special reference to the personal data of the respondents, which will be anonymous. The subjects will be collected at the Osijek Clinical Hospital Center - Clinic for Anesthesiology, Reanimation and Intensive Care at the Institute for Pain Management. Patients who meet the criteria for inclusion in the research will be asked to participate in it and will be explained to them verbally and in writing using the information form for the subjects. After signing the informed consent, patients will be encrypted for data and identity protection.

On the specified day, they will be asked to fill out a questionnaire (ODI, PSQI, SF-36, MCGill short, HAQ, painDETECT), then allow blood sampling, and a physiotherapeutic assessment - mobility range (goniometry), circularity measurements, and Time up and go tests. Sit up test, Adams Forward Bend test, Lasegue test, walk on toes test, walk on heel test and toe-floor distance test. The above physiotherapeutic tests are used in the standard assessment of patients.

Patients will be asked to fill out a questionnaire at the follow-up examination, at the end of therapy and at the next follow-up examination, after 3 months.

The first and control examinations will be performed by a competent doctor, specialist. Blood sampling will be performed according to control at the Osijek Clinical Hospital Center, if the control is not scheduled, and for research purposes it will be performed at the Mursa Medical Center. From the laboratory findings, leukocytes, C-reactive protein (CRP) and differential blood count (DKS) and cytokine levels will be measured.

Blood samples for analysis will be collected in test tubes with red caps, which will be stored at +4 until centrifugation in the Translational Medicine Laboratory of the Faculty of Dental Medicine and Health Osijek. The sample will be centrifuged at 1000 rcf/10min and then the serum will be aliquoted into separate sterile test tubes and stored in a refrigerator at -80°C until laboratory analysis. For multicomplex quantitative analysis of anti-inflammatory cytokines, interferon gamma, tumor necrosis factor alpha, chemokine ligand and matrix metalloproteinases will be used customized ProcartaPlex Multiplex tests (eBioscience, Affymetrix) whose principle is based on beads for protein quantification according to the principle of the Sedwich ELISA test with the use of Luminex® xMAP® (multi -analyte profiling) The entire protocol will be carried out according to the manufacturer's eBioscience instructions. The plate will be read in the Luminex® xMAP® device. The level of the tested analytes will be determined using the ProcartaPlex Analyst v1.0 software. eBioscience, Affymetrix).

To calculate the appropriate number of respondents, statistical methods will be applied as follows: - to observe a medium effect (f = 0.25) in the difference of continuous variables between three measurements in two groups of subjects, the total minimum required sample size is 44 subjects - to observe a medium effect (d = 0.5) in the difference of continuous variables between two groups of subjects, with a significance level of 0.05 and a power of 0.80, the minimum required sample size is 128 subjects. In conclusion, the minimum sample size in the research is 128 respondents (G*Power, 3.1.2).

Numerical data will be described by the arithmetic mean and standard deviation, and in the case of distributions that do not follow a normal distribution, by the median and interquartile range. Differences between two independent groups of normally distributed numerical data will be tested by Student's T-test, in case the variables do not follow a normal distribution, a non-parametric analogue (Man-Whitney U test) will be used. Statistical analysis will be performed with the Statistica 10.0 program (StatSoft, Tulsa, OK, USA), with a selected significance level of α=0.05.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes; age 18-70 years;
* unilateral radicular pain of the lumbar segment;
* diagnosis: intervertebral disc herniation;
* confirmed diagnosis by clinical picture;
* consent to participate in the study, which is confirmed by signing the informed consent;
* unilateral lumbar radicular pain;
* duration of pain up to six months;
* symptomatic disc herniation at one level;
* pain intensity measured by the VAS scale from 0 to 10, which is equal to or greater than 5;
* pain intensity along the leg

Exclusion Criteria:

* patients younger than 18 or older than 70 years;
* refusal of patients to participate in research;
* patients with systemic, local infections in the area of the lumbar spine;
* dermatological diseases in the area of the lumbar spine;
* pregnancy;
* central stenosis of the lumbar canal;
* patients with bilateral radicular pain;
* lumbar radicular pain caused by causes other than a herniated disc;
* allergy to steroids, local anesthetics, fentanyl, midazolam and contrast media;
* positive history of prolonged bleeding;
* local or systemic infection; previous lumbar spine surgery;
* abuse of opioids;
* proven inflammatory rheumatic disease;
* proven inflammatory bowel disease;
* other infections.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2024-09-02 (Actual); Primary Completion 2026-03-02 (Estimated); Study Completion 2026-03-02 (Estimated)

PRIMARY OUTCOMES:
Using standard biochemical analyses, measure the concentrations of pro-inflammatory and anti-inflammatory cytokines and metallopeptidases in the serum before physical therapy, i.e. ESI, and two weeks and three months after the start of said therapies. | Up to 3 months
  There will be changes in the concentrations of pro-inflammatory and anti-inflammatory cytokines and matopeptidases in the serum, like interleukin 1β (IL-1β), interleukin 6 (IL-6), interleukin 8 (IL-8), interferon gamma (INF-γ), tumor necrosis factor alpha or gamma (TNF-α), chemokine ligand 3 (CCL3) and matrix metalloproteinases MMP-3 and MMP-9, during physical therapy, that is, the minimally invasive application of epidural steroid injection therapy in patients with pain caused by the bulging of the intervertebral disc in the lumbar part of the spine, and whether these changes are expressed when using both methods.

SECONDARY OUTCOMES:
Determine the degree of the patient's psychophysical condition and quality of life | Up to 3 months
  Physical therapy, i.e. therapy with epidural steroid injection on possible changes in the clinical status, psychophysical function and quality of life of patients with questionnaire: For pain-Visual Analogue Pain Scale (VAS), McGill short and painDETECT. The questionnaires for the percentage of disability, physical functioning,health status and quality of life - Oswestry low back pain disability questionnaire (ODI), 36-Item Short Form Survey (SF-36) and Health Assessment Questionnaire (HAQ). Pittsburgh Sleep Quality Index (PSQI) - for sleep quality, sleep disturbances and use of sleep medications. With these questionnaires I want to establish whether changes in these parameters are reflected in changes in the concentrations of pro-inflammatory or anti-inflammatory cytokines and metallopeptidases in order to possibly identify new biological markers that would could be used in monitoring the outcome of treatment when applying physical therapy, that is, ESI.

CONTACTS AND LOCATIONS:
Overall Officials: Karla Rožac, Master's, Principal Investigator — Faculty of Dental Medicine and Health Osijek
Locations (1):
- Faculty of Dental Medicine and Health Osijek, Osijek, Croatia

IPD SHARING:
Plan to Share IPD: No
I do not plan to make IPD available to other researchers. IPDs will be administrated and stored by one person.

REFERENCES:
- [Background] Budrovac D, Rados I, Hnatesen D, Harsanji-Drenjancevic I, Tot OK, Katic F, Lukic I, Skiljic S, Neskovic N, Dimitrijevic I. Effectiveness of Epidural Steroid Injection Depending on Discoradicular Contact: A Prospective Randomized Trial. Int J Environ Res Public Health. 2023 Feb 19;20(4):3672. doi: 10.3390/ijerph20043672. PMID 36834367